CLINICAL TRIAL: NCT00401947
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Multiple Doses of ACH-0137171 in Subjects With Chronic Hepatitis C Infection
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of ACH-0137171 in Participants With Chronic Hepatitis C Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Nephrotoxicity
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Achillion, a wholly owned subsidiary of Alexion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ACH171-002
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: HCV Infection
Keywords: HCV; Chronic; Hepatitis
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome; Hepatitis

INTERVENTIONS:
Drug: ACH-0137171

SUMMARY:
The purpose of this study was to investigate the safety, tolerability, pharmacokinetics (PK), and antiviral activity of multiple doses of ACH-0137171 in participants with chronic hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, dose-escalation study of ACH-0137171 in participants with chronic HCV infection.

Sequential cohorts of 10 participants were randomized (8:2) to receive multiple doses of ACH-0137171 or placebo for 4 days (Days 1 through 4) with a single dose on Day 5 followed by a complete PK profile. Dosing was 300-600 milligrams (mg) administered either every 12 hours or every 6 hours (maximum daily dose of 2400 mg). All doses were administered with food.

The dose cohorts were as follows:

Study Schema:

Cohort 1: 300 mg ACH-0137171/placebo every 12 hours (600 mg/day) Cohort 2: 300 mg ACH-0137171/placebo every 6 hours (1200 mg/day) Cohort 3: 600 mg ACH-0137171/placebo every 6 hours (2400 mg/day)

A full review of all safety data will occur following each cohort. Depending on the data, the Sponsor, in consultation with the Principal Investigator(s), may consider modifying the planned dose escalation. The Sponsor may choose to interject an intermediate dose cohort between 2 planned dose escalations or repeat a given dose level, or extend the dosing period, or add an additional cohort. If a similar Grade 3 or 4 adverse event occurs in 3 or more participants and was considered to be at least possibly related to the study drug, escalation to a higher dose will not occur.

Serial HCV ribonucleic acid (RNA) measurements, PK measurements of plasma concentrations of ACH-0137171, and periodic safety monitoring occurred on Days 1 through 5. Additional HCV RNA and PK measurements were taken on Days 6 through 9. Follow-up safety evaluations will be completed 14 days after the last study drug administration (that is, on Days 12 and 19).

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection must be documented by positive anti-HCV antibody using a third-generation enzyme immunoassay and persistent detection of HCV RNA in the blood for at least 6 months.
* Participants must be infected with HCV genotype 1 (line probe assay; INNO-LiPA HCV II, Innogenetics) and maybe treatment-naïve or treatment-experienced (treatment experienced specifically means prior treatment with interferon, standard or pegylated, with or without ribavirin with therapy stopped > 6 months prior to screening).
* Eligible participants must have had alanine aminotransferase and aspartate aminotransferase < 5 x upper limit of normal (ULN), plasma HCV RNA > 5 log10 international units (IU)/milliliter (mL), and have had no clinical or laboratory evidence of hepatic decompensation for inclusion (must have platelets > 100,000/cubic millimeter [mm^3], total bilirubin < 1.5 x ULN, prothrombin time < 1.5 x ULN, or albumin > 3.0 grams/deciliter [g/dL] for inclusion).
* Women were eligible if not pregnant or breast-feeding.
* Women of childbearing potential (that is, not surgically sterile or confirmed post menopausal) must have had confirmed negative pregnancy tests. All participants must practice a medically acceptable form of contraception.

Exclusion Criteria:

* Human immunodeficiency virus or hepatitis B virus co-infection known cirrhosis.
* Prior history of clinical hepatic decompensation (ascites, jaundice, encephalopathy, or variceal hemorrhage), alcoholic or other forms of chronic liver disease, evidence of hepatocellular carcinoma (α-fetoprotein > 50 nanograms/mL), creatinine clearance < 80 mL/minute (using Cockcroft-Gault equation), hemoglobin < 10 g/dL, neutrophils < 1500/mm^3, and abnormal thyroid function tests (thyroid stimulating hormone > 2.5 microIU/mL, free T4 > ULN), or, a positive test result for illicit drugs, alcohol, or drug abuse within the past 12 months.
* Participants who have had significant gastrointestinal, thyroid, renal, cardiovascular, pulmonary, oncologic, or neurological disease, or who are currently receiving immunomodulators (corticosteroids), investigational, nephrotoxic or hepatotoxic drugs (for example, phenytoin, carbamazepine, isonicotinic acid hydrazide, azole anti-fungal agents such as ketoconazole, and aminoglycoside antibiotics), non-steroidal anti-inflammatory agents, ibuprofen or acetaminophen (on a daily basis) will also be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-11-30 (Actual); Study Completion 2007-03-31 (Actual)

PRIMARY OUTCOMES:
To assess the short-term safety and tolerability of multiple, escalating, oral doses of ACH-0137171 in subjects with chronic hepatitis C infection.
To characterize the plasma pharmacokinetics of ACH-0137171 following administration of multiple, escalating, oral doses in subjects with chronic hepatitis C infection.
To assess the antiviral activity of ACH-0137171 as measured by plasma HCV RNA levels in subjects with chronic hepatitis C infection following administration of multiple, escalating, oral doses.
To assess the correlation between antiviral activity and pharmacokinetic parameters.

SECONDARY OUTCOMES:
To perform viral dynamic and pharmacodynamic modeling of ACH 0137171 virologic response.
To assess the biochemical response of ACH-0137171 as measured by the change from baseline of serum ALT and AST levels.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, San Antonio, Texas
- Clinical Trial Site, Berlin, Germany
- Clinical Trial Site, Utrecht, Netherlands